CLINICAL TRIAL: NCT03060928
Title: Evaluation of Tendon-to-Bone Healing Potential in Arthroscopic Rotator Cuff Repair Through Biological Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Roberto Leo, MD, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 753_2016
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Artelon®
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — polyetherurethane urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Arthroscopic Rotator Cuff Repair with standard treatment
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair
- Experimental 1 (Experimental): Arthroscopic Rotator Cuff Repair with standard treatment + biological stimulation with micro-perforations
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair; Procedure: Micro-perforations
- Experimental 2 (Experimental): Arthroscopic Rotator Cuff Repair with standard treatment + biological stimulation with the combination of micro-perforations and use of Artelon® Tissue Reinforcement
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair; Procedure: Micro-perforations; Procedure: Artelon®

INTERVENTIONS:
Procedure: Arthroscopic Rotator Cuff Repair — Arthroscopic Rotator Cuff Repair
Procedure: Micro-perforations — Biological stimulation with micro-perforations
  Arms: Experimental 1; Experimental 2
Procedure: Artelon® — Biological stimulation with Artelon® Tissue Reinforcement
  Arms: Experimental 2

SUMMARY:
Evaluation of clinical and radiological outcomes in patients undergoing Arthroscopic Rotator Cuff Repair with standard treatment compared to patients receiving biological stimulation with micro-perforations or with the combination of micro-perforations and use of Artelon® Tissue Reinforcement, a synthetic device based on degradable polyurethaneurea.

The investigators believe that this kind of tendon-to-bone healing stimulation with the two proposed methods can increase the repair quality by significantly decreasing the lesion recurrence rate (currently described for 15% of patients) and can improve various parameters such as pain, range of motion and strength, thereby hastening the return to daily activities and psycho-physical well-being.

ELIGIBILITY:
Inclusion Criteria:

* a medium rotator cuff tear (from 1 to 3 cm, according to Cofield Classification) with an indication for arthroscopic repair
* signed informed consensus

Exclusion Criteria:

* previous fractures
* diabetes
* subscapularis tears
* tears < 1cm or > 3 cm
* reduced passive range of motion
* infections
* known mental or neurological disorders unwilling or unable to follow the post-surgery instructions
* conditions that contraindicate arthroscopic rotator cuff surgery
* patients without complete osteogenesis
* pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Retear rate | 12 months post-operatively
  Comparison of re-ruptures rate in each group evaluated with magnetic resonance imaging

SECONDARY OUTCOMES:
Constant-Murley | 3, 6, 12 months post-operatively
  Comparison of Constant-Murley Score in each group
DASH | 1, 3, 6, 12 months post-operatively
  Comparison of DASH Score in each group
VAS | 1, 3, 6, 12 months post-operatively
  Comparison of Visual Analogue Scale (VAS) in each group
Passive ROM | 1, 3, 6, 12 months post-operatively
  Comparison of passive range of motion in each group
Adverse events | 1, 3, 6, 12 months post-operatively
  Adverse events for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Leo, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided